CLINICAL TRIAL: NCT05632146
Title: COMPARISON OF CONTINUOUS VERSUS INTERRUPTED-X SUTURING TECHNIQUE FOR CLOSURE OF RECTUS SHEATH IN PATIENTS UNDERGOING EMERGENCY LAPAROTOMY FOR HOLLOW VISCUS PERFORATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KingEdwardMU1
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Duodenal Perforation; Bowel Perforated
MeSH Terms: conditions — Intestinal Perforation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with hollow viscus perforation (Active Comparator)
  Interventions: Procedure: Continuous suturing; Procedure: Interrupted X suturing
- Patient with hollow viscus perforation (Active Comparator)
  Interventions: Procedure: Continuous suturing; Procedure: Interrupted X suturing

INTERVENTIONS:
Procedure: Continuous suturing — In continuous closure, each bite will be taken 2 cm from the cut edge of linea alba and successive bites taken 1 cm from each other in continuous fashion followed by gentle approximation of the wound
Procedure: Interrupted X suturing — In interrupted X closure, large bite will be taken outside-in, 2 cm from the cut edge of linea alba and the needle emerged on the other side from inside out diagonally 2 cm from the edge and 4 cm below the first bite and this strand will be crossed and continued outside-in, diagonally at 90 degree to the first diagonal. The two ends will be tied just tight enough to approximate the edges of linea alba.

SUMMARY:
THIS STUDY IS GOING TO COMPARE THE INCIDENCE OF BURST ABDOMEN IN PATIENTS UNDERGOING LAPAROTOMY WOUND CLOSURE IN CONTINUOUS VERSUS INTERRRUPTED-X MANNER

DETAILED DESCRIPTION:
An emergency laparotomy is a common surgical procedure, performed for a wide variety of intra-abdominal pathologies, which has a significant associated morbidity and mortality. Each year, approximately 30,000 emergency laparotomies are performed in the UK [1]. A major surgical complication after emergency midline laparotomy is abdominal fascial dehiscence. Dehiscence is associated with increased morbidity and mortality rates up to 30%, prolonged hospital stay, and a long-term risk of developing incisional hernia [1].

Hollow viscus perforation is one of the most common cause of peritonitis necessitating emergency surgical intervention. The diagnosis is mainly based on clinical grounds. Plain abdominal X-rays (erect) may reveal dilated and edematous intestines with pneumoperitoneum. Local findings include abdominal tenderness, guarding or rigidity, distension, diminished bowel sounds and systemic findings include fever, chills or rigor, tachycardia, sweating, tachypnea, restlessness, dehydration, oliguria, disorientation and ultimately shock. Exposure of the normally sterile peritoneal cavity to intraluminal contents causes secondary bacterial peritonitis. The peritoneal contamination due to bowel perforation is one of the leading risk factor for occurrence of burst abdomen [2].

Laparotomy wound dehiscence (LWD) is a term used to describe separation of the layers of a laparotomy wound before complete healing has taken place. Other terms used interchangeably are acute laparotomy wound failure and burst abdomen. Frequency of laparotomy wound dehiscence in the relevant literature is cited in the range of 0.2% to 10%[3,4]. The occurrence of fascial dehiscence represents a risk factor for increased mortality rates of up to 25%[5] Acute wound failure may be occult or overt, partial or complete. Overt wound failure follows early removal of sutures leading to evisceration. Occult dehiscence occurs with disruption of musculo-aponeurotic layer beneath intact skin sutures. Wound dehiscence has been noted to occur when a wound fails to gain sufficient strength to withstand stresses placed upon it. The separation may occur when overwhelming forces break sutures, when absorbable sutures dissolve too quickly or when tight sutures cut through tissues [6].

Conventional continuous closure technique has been shown to compromise blood supply and thereby poor wound holding, during initial phases of wound dehiscence. Surgeons have been continuously striving to overcome postoperative complications associated with laparotomy wound closure using newer techniques and newer suture materials. Several reviews have studied the optimal suture repair for closing the abdominal fascia, but no consensus has been reached. Hence, it is imperative for us to ascertain better method of closing the abdomen. While the choice may not be so important in elective patients who are nutritionally adequate, do not have any risk factor for dehiscence and are well prepared for surgery, however it may prove crucial in emergency patients who often have multiple risk factors for developing dehiscence and the strangulation of the sheath is the proverbial last straw in precipitating wound failure [7].

A number of studies have been conducted which suggest that new interrupted X-technique for abdominal closure after midline laparotomy significantly reduces the risk of burst abdomen [8,9]. A study done by Balaji C et al comparing continuous versus interrupted X suture technique showed that incidence of wound dehiscence was 10 % in patients who underwent interrupted X closure and 36% in patients who underwent continuous closure [10]. However, these studies haven't taken into account a specific study population with similar pathology and risk of burst abdomen to compare the two suturing techniques. So, the aim of the present study is to compare the prevalence of burst abdomen in patients undergoing midline abdominal wall closure with interrupted X-suturing technique and continuous suturing technique in patients with enteric perforation.

ELIGIBILITY:
Inclusion Criteria:

* All patients of both genders with age greater than 18 years, undergoing emergency laparotomy through midline incision for hollow viscus perforation.
* ASA grade III

Exclusion Criteria:

* Patients who had undergone a previous laparotomy for any condition or had an incisional hernia or burst abdomen at presentation.
* Patients undergoing laparotomy with anterior abdominal wall injury in the form of muscle hematoma, disruption or abdominal wall laceration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-11-03 (Estimated)

PRIMARY OUTCOMES:
Burst abdomen | 1-14 days
  It is defined as partial or complete separation of the abdominal musculo-aponeurotic layer leading to protrusion or evisceration of abdominal contents.

SECONDARY OUTCOMES:
Pain score | 1-14 days
  Pain score will be assessed post-operatively using visual analogue score ranging from 0 to 10 with 0 being no pain and 10 being the worst pain
Superficial surgical site infection | 1-14 days
  Pain, tenderness, localized swelling, erythema at wound site and surgeon open up the superficial incision, revealing purulent discharge and confirmation of pathogen on culture grown from aseptically harvested wound discharge.
Deep surgical site infection | 1-14 days
  Infection within peritoneal cavity presenting with purulent discharge from a drain with pathogen confirmed on culture or abdominal collection documented on USG will be labelled as deep surgical site infection.

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University / Mayo Hospital, Lahore, Punjab Province, Pakistan